CLINICAL TRIAL: NCT02311907
Title: The Use of Glutathione (GSH) for Prevention of Paclitaxel/Carboplatin (TAXOL/CBDCA) Induced Peripheral Neuropathy: A Phase III Randomized, Double-Blind Placebo Controlled Study
Brief Title: Glutathione in Preventing Peripheral Neuropathy Caused by Paclitaxel and Carboplatin in Patients With Ovarian Cancer, Fallopian Tube Cancer, and/or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: N08CA; NCI-2011-01965 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000654097; U10CA037404 (NIH); NCT00979082 (obsolete NCT alias)
Record Dates: First submitted 2014-12-08; First posted 2014-12-09 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Chemotherapeutic Agent Toxicity; Neuropathy; Neurotoxicity Syndrome; Pain; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Glutathione; Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (glutathione, carboplatin) (Experimental): Patients receive glutathione intravenously (IV) over 15 minutes, paclitaxel* IV over 1 or 3 hours depending on planned dose cycle length and carboplatin IV over 30 minutes.
  Interventions: Drug: Carboplatin; Drug: Glutathione; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm II (placebo, paclitaxel) (Placebo Comparator): Patients receive placebo IV over 15 minutes, paclitaxel* IV over 1 or 3 hours depending on planned dose cycle length and carboplatin IV over 30 minutes.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Carboplatin — Given IV, over 30 minutes per planned chemotherapy regimen
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Glutathione — Given IV, over 15 minutes, immediately before chemotherapy administration
  Other Names: Glutham; GSH; Reduced Glutathione
  Arms: Arm I (glutathione, carboplatin)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV, over 1 or 3 hours, per planned chemotherapy regimen
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo, paclitaxel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial is studying glutathione to see how well it works in preventing peripheral neuropathy caused by paclitaxel and carboplatin in patients with ovarian cancer, fallopian tube cancer, and/or primary peritoneal cancer. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Chemoprotective drugs, such as glutathione, may help prevent peripheral neuropathy caused by paclitaxel and carboplatin. It is not yet known whether glutathione is more effective than a placebo in preventing peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare TAXOL (paclitaxel)/carboplatin (CBDCA) induced peripheral neuropathy as measured by European Organization for Research and Treatment of Cancer (EORTC)- Quality of Life (QOL)-chemotherapy induced peripheral neuropathy 20 (CIPN20) between glutathione (GSH) and placebo arms.

SECONDARY OBJECTIVES:

I. To compare the incidences of grade 2+ and grade 3+ TAXOL/CBDCA induced peripheral neuropathy measured by Common Terminology Criteria for Adverse Events (CTCAE) neuropathy scale between GSH and placebo arms.

II. To compare the time to onset of grade 2+ and grade 3+ TAXOL/CBDCA induced peripheral neuropathy between GSH and placebo arms, measured by CTCAE neuropathy scale.

III. To compare the proportion of patients requiring chemotherapy dose reductions secondary to TAXOL/CBDCA induced peripheral neuropathy between GSH and placebo arms.

IV. To compare the proportion of patients stopping TAXOL/CBDCA secondary to peripheral neuropathy between GSH and placebo arms.

V. To assess the toxicity profile of GSH in this situation. VI. To evaluate whether GSH influences the anti-tumor activity of TAXOL/CBDCA. VII. To evaluate patient quality of life (QOL) measured by Functional Assessment of Cancer Therapy-Ovarian (FACT-O) (ovarian/fallopian tube/primary peritoneal cancer patients only) and patient daily symptom questionnaires over time between GSH and placebo arms.

TERTIARY:

I. To explore the association of genetic variations in genes involved in taxane/platinum metabolism with incidence of grade 2+ TAXOL/CBDCA induced peripheral neuropathy.

II. As part of ongoing research for North Central Cancer Treatment Group (NCCTG) studies, we are banking blood products for future studies.

OUTLINE:

Patients are stratified according to baseline neuropathy (none vs grade 1), debulked status (no gross residual disease [no clinically apparent residual lesions at the completion of primary surgery] vs optimal [largest residual lesion < 1 cm at primary surgery] vs sub-optimally debulked [residual lesion > 1 cm] or not operated upon), and cancer type (ovarian/fallopian tube/primary peritoneal cancers vs lung cancer vs other). Patients are randomized to 1 of 2 treatment arms. Patients are grouped based on, Planned paclitaxel dose cycle length (Weekly vs. every 3 weeks vs. every 4 weeks). The stratification factors listed include demographic, prognostic factors and medication that can potentially impact the primary or secondary outcomes, so they need to be distributed evenly among the two arms. The 18 level combinations involved in these four stratification factors are within the maximum recommended of one half of the group sample size for the study.

Ideally, patients begin receiving glutathione before their first dose of chemotherapy, but must begin glutathione before their second dose of chemotherapy.

ARM I: Patients receive glutathione intravenously (IV) over 15 minutes, paclitaxel* IV over 1 or 3 hours depending on planned dose cycle length and carboplatin IV over 30 minutes.

ARM II: Patients receive placebo IV over 15 minutes, paclitaxel* IV over 1 or 3 hours depending on planned dose cycle length and carboplatin IV over 30 minutes.

NOTE: *Alternatively, patients may receive paclitaxel IV over 1 hour and glutathione/placebo IV over 15 minutes weekly and carboplatin every 21 days for 12 weeks.

Blood samples are collected periodically for pharmacogenomic and other biomarker analyses. Patients complete questionnaires periodically, including quality-of-life assessments.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo treatment with TAXOL at 150-200 mg/m2 and CBDCA at area under the curve (AUC) = 5-7 every 21 or 28 days for at least 12 weeks; alternatively, paclitaxel can be prescribed at 80 mg/m2 weekly for at least 12 weeks, with the same CBDCA dose of AUC = 5-7 every 21 days; additional chemotherapy agents are allowed (bevacizumab, etoposide, etc) per physician discretion, as long as they are not known to be neurotoxic; Note: patients ideally will begin GSH therapy prior to their first dose of this chemotherapy, but must begin GSH therapy prior to their second dose of chemotherapy
* Ability to sign informed consent and understand the nature of a placebo-controlled trial
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to complete English language questionnaire(s) by themselves or with assistance
* Life expectancy >= 6 months
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only, per clinician discretion
* Willingness to provide blood specimens as required by the protocol
* White blood cell (WBC) >= 3400
* Absolute neutrophil count (ANC) >= 1500
* Platelet (PLT) >= 100,000
* Hemoglobin (HgB) > 10.0
* Creatinine =< 1.5 x upper limit of normal (ULN)

Exclusion Criteria:

* Pre-existing history of peripheral neuropathy > grade 1 (National Cancer Institute [NCI] CTCAE version [v] 4.0) due to any cause (e.g., chemotherapy, diabetes, alcohol, toxin, or heredity)
* Other medical conditions, which in the opinion of the treating physician/allied health professional would make this protocol unreasonably hazardous for the patient
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Prior TAXOL and/or CBDCA chemotherapy treatment (other than the current treatment regimen)
* Concurrent use of any agent being used specifically to prevent or treat neuropathy, including but not limited to the following:

  * Gabapentin
  * Glutamine powder or glutamine tablets
  * Vitamin B6 or E

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (390):
- United States (390):
  - Providence Hospital, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Northbay Cancer Center, Fairfield, California
  - Cancer Care Associates of Fresno Medical Group Inc, Fresno, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Feather River Cancer Center, Paradise, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan St. Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Louisiana State University Sciences Center- Monroe, Monroe, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - The Memorial Hospital at Easton, Easton, Maryland
  - Cancer Trials Support Unit, Rockville, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - McLaren-Macomb, Mount Clemens, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Glens Falls Hospital, Glens Falls, New York
  - Staten Island University Hospital, Staten Island, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson AFB, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Cancer Centers of the Carolinas-Greer Medical Oncology, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford NCI Community Oncology Research Program of the North Central Plains, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 195 patients were enrolled, 185 started the treatment (8 cancels, 1 ineligible and 1 excluded due to switching regimens).
Groups:
- A (Glutathione, Carboplatin): Patients receive glutathione IV over 15 minutes, paclitaxel* IV over 3 hours, and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21-28 days for at least 12 weeks in the absence of disease progression or unacceptable toxicity.
- B (Placebo, Paclitaxel): Patients receive placebo IV over 15 minutes, paclitaxel* IV over 3 hours, and carboplatin IV over 30 minutes as in arm A.
Period: Overall Study
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Started | 94 | 91
Completed | 94 | 91
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel) | Total
Number analyzed (Participants) | 94 | 91 | 185
Age, Continuous [Median (Full Range); unit: years] | 63 [37 to 85] | 63 [28 to 84] | 63 [28 to 85]
Gender [Count of Participants; unit: Participants]
  Female | 74 | 76 | 150
  Male | 20 | 15 | 35
Region of Enrollment [Number; unit: participants]
  United States | 94 | 91 | 185

OUTCOME MEASURES:

1. Primary Outcome: Paclitaxel/Carboplatin (PC) Induced Peripheral Neuropathy as Assessed by EORTC QLQ-CIPN20 (European Organization for Research and Treatment of Cancer (EORTC), Quality of Life (QLQ), Chemotherapy Induced Peripheral Neuropathy 20 (CIPN20)).
Description: The CIPN sensory subscale will be calculated by standard scoring algorithm and converted to 0-100 scale (higher scores indicated less symptoms and better quality of life). Generalized linear models (repeated measures analysis of variance [ANOVA] if data are complete) will be used to compare the CIPN between Glutathione (GSH) and placebo arms.
Time Frame: Every 28 day cycle, up to 6 cycles.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale 1-100
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 94 | 91
Units on a scale 1-100 | 83.7 (0.89) | 82.1 (0.93)
Statistical Analysis 1: Comparison: A (Glutathione, Carboplatin) vs B (Placebo, Paclitaxel); Generalized linear models (repeated measures analysis of variance [ANOVA]) will be used to compare the CIPN between GSH and placebo arms; Test type: Superiority or Other; p = 0.21, ANOVA

2. Secondary Outcome: Recurrence-free Survival (for Patients Without Clinical Evidence of Disease)
Description: A log-rank test and a Kaplan-Meier curve will be used to compare the recurrence free survival between GSH and placebo arms (for ovarian/fallopian tube/primary peritoneal patients only).
Time Frame: Up to 1 year
Population: Patients without clinical evidence of disease.
Measure: Median (95% Confidence Interval); unit: Median survival time in days
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 45 | 40
Median survival time in days | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: A (Glutathione, Carboplatin) vs B (Placebo, Paclitaxel); Test type: Superiority or Other; p = 0.63, Log Rank

3. Secondary Outcome: Change in Patient Reported Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Ovarian (FACT-O) and Patient Daily-symptom Questionnaires Over Time.
Description: Quality of life was measured by FACT-O (on a 0 to 100 scale, higher scores represent better life quality) from baseline and at the end of TAXOL/CBDCA. The change in Quality of Life was calculated as the difference between baseline measure and end of treatment measure (with range from -100 to 100). A negative change represents a worsening in QOL from baseline to one year. Abbreviations used: Change from Baseline (chg from bsl)
Time Frame: Baseline to 1 year
Population: FACT-O Change from Baseline to cycle 6 data available for 34 patients.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 17 | 17
units on a scale
  FACT-O Physical Subscale Chg from Bsl | -14.3 [-57.1 to 57.1] | -8.9 [-75.0 to 14.3]
  FACT-O Social/Family Subscale Chg from Bsl | -4.2 [-28.6 to 4.2] | 0.0 [-100.0 to 21.4]
  FACT-O Emotional Subscale Chg from Bsl | 8.3 [-45.8 to 37.5] | 4.2 [-20.8 to 45.8]
  FACT-O Functional Subscale Chg from Bsl | 0.0 [-32.1 to 21.4] | 5.1 [-96.4 to 42.9]
  FACT-O Additional Concerns Subscale Chg from Bsl | -2.3 [-22.7 to 20.5] | 4.8 [-29.5 to 19.8]
  FACT-O Total Score Chg from Bsl | 0.3 [-27.6 to 13.3] | 4.4 [-39.5 to 16.1]

4. Secondary Outcome: Paclitaxel Acute Pain Syndrome Incidence and Severity Between GSH and Placebo Arms
Description: Descriptive statistics will be used to describe TAXOL/CBDCA acute pain syndrome incidence/severity between GSH and placebo arms. Pain was scored on a scale from 0-10, where 0 = 'No aches or pains' and 10 = 'Aches or pains as bad as can be.'
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: units on a scale
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 94 | 91
units on a scale | 2.0 [0 to 10] | 2.0 [0 to 10]

5. Secondary Outcome: Percentage of Patients Delaying PC Chemotherapy Secondary to PN
Description: Patients delaying TAXOL/CBDCA secondary to peripheral neuropathy between GSH and placebo arms.
Time Frame: Up to 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 94 | 91
Percentage of participants | 1.1 | 0

6. Secondary Outcome: Percentage of Patients Undergoing Dose Reductions Secondary to PCI PN
Description: Proportion of patients requiring chemotherapy dose reductions secondary to TAXOL/CBDCA induced peripheral neuropathy between GSH and placebo arms.
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 94 | 91
percentage of participants
  Reduced TAXOL Dose : Yes | 2.1 | 1.1
  Reduced CARBO Dose: Yes | 1.1 | 0.0

7. Secondary Outcome: Percentage of Patients With Grade 2+ and Grade 3+ Paclitaxel/Carboplatin-induced (PCI) Peripheral Neuropathy (PN) According to the Common Terminology Criteria for Adverse Events (CTCAE) Neuropathy Scale
Description: Proportion of grade 2+ and grade 3+ chemotherapy induced peripheral neuropathy (CIPN) at any time during or at the end of the TAXOL/CBDCA based chemotherapy between GSH and placebo arms. Neuropathy scale has grades 1 through 5 (1-mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening and Grade 5 Death related to AE).
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 94 | 91
percentage of participants
  Grade 2+ CIPN: Yes | 38.3 | 33.0
  Grade 3+ CIPN: Yes | 5.3 | 4.4

8. Secondary Outcome: Times to Onset of CTCAE Grade 2+ PN
Description: Compare time to grade 2+ CIPN between GSH and placebo arms.
Time Frame: Up to 1 year
Population: Number of Participants analyzed is 93 for Arm I due to error in date entered.
Measure: Median (Standard Error); unit: days
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 93 | 91
days | 140 (18.5) | 234 (26.1)

9. Secondary Outcome: Times to Onset of CTCAE Grade 3+ PN
Description: Time to grade 3+ CIPN between GSH and placebo arms.
Time Frame: Up to 5 years from registration
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Number analyzed (Participants) | 94 | 91
days | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

ADVERSE EVENTS:
Groups:
- A (Glutathione, Carboplatin); B (Placebo, Paclitaxel): Quality-of-Life Assessment: Ancillary studies
Arm/Group | A (Glutathione, Carboplatin) | B (Placebo, Paclitaxel)
Serious Adverse Events (participants affected / at risk) | 7/94 | 1/91
Other Adverse Events (participants affected / at risk) | 64/94 | 62/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (Glutathione, Carboplatin) (N=94) | B (Placebo, Paclitaxel) (N=91)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (Glutathione, Carboplatin) (N=94) | B (Placebo, Paclitaxel) (N=91)
Anemia (Blood and lymphatic system disorders) | 12 (22) | 15 (28)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Death NOS (General disorders) | 3 (3) | 2 (3)
Edema limbs (General disorders) | 2 (3) | 0 (0)
Edema trunk (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 10 (18) | 9 (11)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2)
Anaphylaxis (Immune system disorders) | 2 (2) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (3) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (3) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative ocular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1) | 1 (1)
INR increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (5) | 7 (15)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 22 (44) | 17 (31)
Platelet count decreased (Investigations) | 6 (8) | 10 (18)
Weight gain (Investigations) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 9 (13) | 9 (14)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (7) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6) | 5 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (20) | 7 (12)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (11) | 4 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 6 (7)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 5 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes